CLINICAL TRIAL: NCT05809687
Title: Evaluate Efficacy and Safety of DKP21102_B Added on to DKP21102_A Compared With DKP21102_A in Mixed Dyslipidemia Patients
Brief Title: Phase 3 Trial to Evaluate the Efficacy and Safety of DKP21102_B Added on to DKP21102_A Compared With DKP21102_A
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The clinical trial was withdrawn due to a commercial decision.
Sponsor: Dongkwang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DKP21102_301
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-09

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): DKP21102_A, DKP21102_C
  Interventions: Drug: DKP21102_C; Drug: DKP21102_A
- Treatment group (Experimental): DKP21102_A, DKP21102_B
  Interventions: Drug: DKP21102_B; Drug: DKP21102_A

INTERVENTIONS:
Drug: DKP21102_C — Placebo
  Arms: Control group
Drug: DKP21102_B — Treatment
  Arms: Treatment group
Drug: DKP21102_A — Active Control

SUMMARY:
Phase 3 study to evaluate the efficacy and safety of DKP21102_B Added on to DKP21102_A Compared with DKP21102_A

DETAILED DESCRIPTION:
Phase 3 study to evaluate the efficacy and safety of DKP21102 in patients with mixed dyslipidemia where LDL-C is properly controlled but triglyceride and HDL-C levels are not regulated by DKP21102_A alone.

ELIGIBILITY:
Inclusion Criteria:

* A man or woman over 19 years old.
* Patients with coronary heart disease or risk of coronary heart disease

Exclusion Criteria:

* History of Unstable angina, myocardial infarction etc
* Uncontrolled hypo-thyroidism (TSH≥1.5XULN), Diabetes(HbA1c ≥ 9.0%)
* renal impairment (Creatinine clearance < 60 mL/min) etc.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent change (%) of non-HDL-C from baseline | from baseline at 12weeks
  non-HDL-C

IPD SHARING:
Plan to Share IPD: No